CLINICAL TRIAL: NCT00776464
Title: Treating Onychomychosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nomir Medical Technologies (Industry)
Responsible Party: nomir medical, Nomir Medical Technologies
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #10-001
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

INTERVENTIONS:
Device: Noveon laser — Two wavelenghts of light

SUMMARY:
A study to treat 4 toes at a time to eliminate Onychomycosis

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* positive onychomycosis
* negative pregnancy

Exclusion Criteria:

* peripheral neuropathy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Complete or near complete disappearance of toenail fungus | 360 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nomir Medical, Waltham, Massachusetts, United States